CLINICAL TRIAL: NCT01335412
Title: Active Surveillance for Adverse Events After Immunization With IXIARO(R) Among U.S. Military Service Personnel
Brief Title: Safety Surveillance After Immunization With IXIARO
Status: Completed | Type: Observational
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: IC51-401
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IXIARO exposed group: Male and female active duty U.S. military personnel ≥ 17 years of age who either received at least one dose of IXIARO
  Interventions: Biological: Japanese Encephalitis Virus vaccine, inactivated, adsorbed
- Comparison group: Male and female active duty U.S. military personnel ≥ 17 years of age who either received at least one dose of JE-VAX

INTERVENTIONS:
Biological: Japanese Encephalitis Virus vaccine, inactivated, adsorbed — 2 x 6mcg / 0.5mL intramuscular injection, Day 0 and 28 (Primary series) or 1x 6mcg / 0.5mL intramuscular injection (Booster)
  Other Names: IXIARO
  Groups: IXIARO exposed group

SUMMARY:
This is an active electronic surveillance using data from the Defense Medical Surveillance System (DMSS) to detect and characterize serious, rare adverse events occurring within 42 days after vaccination with the Japanese Encephalitis Vaccine IXIARO within the US Military, to detect adverse events that occur more frequently after IXIARO and to electronically follow up pregnancies during or shortly before which IXIARO was administered.

There will be no intervention and no individuals contacted.

ELIGIBILITY:
Inclusion Criteria:

* Male and female active duty U.S. military personnel ≥ 17 years of age who either received at least one dose of IXIARO (IXIARO exposed group) or at least one dose of JE-VAX (comparison group).

Exclusion Criteria:

* Individuals who have an ICD-9-CM code suggestive of one of the predefined adverse events screened for in IC51-401 prior to vaccination with IXIARO cannot with certainty be classified as being "disease free" at study entry and will be excluded for that adverse event.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Active duty military personnel (Army, Navy, Air Force, and Marines) who are ≥17 years of age and received at least one dose of Japanese encephalitis vaccine.
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pre-defined, serious adverse events | 42 days after each dose of IXIARO

SECONDARY OUTCOMES:
Detection of non-predefined Adverse Events overrepresented after IXIARO | 42 days after each dose of IXIARO
  Data-mining for overrepresented Adverse events in the IXIARO exposed group compared to comparison group
Occurrence of complications during pregnancy | Up to delivery
  Detect and describe pregnancy complications following inadvertent vaccination in pregnant women
Occurrance of infant health complications | up to 3 months after birth
  Detect and describe infant health complications following inadvertent vaccination in pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Katrin L Dubischar-Kastner, MSc, Study Director — Valneva Austria GmbH
Locations (1):
- Military Vaccine Agency, Alexandria, Virginia, United States